CLINICAL TRIAL: NCT02050646
Title: The Role of Sodium Chloride and the Treg/Th17 Axis in Autoimmune Hepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1303011696; YSOM Pediatrics Department (Other: Yale University School of Medicine)
Record Dates: First submitted 2013-11-04; First posted 2014-01-31 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Autoimmune Hepatitis
Keywords: Autoimmune hepatitis; Liver dysfunction; Elevated serum auto antibodies
MeSH Terms: conditions — Hepatitis, Autoimmune; Liver Diseases | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low salt/ Liberal salt Diet (Experimental): Cross-over trial of liberal salt and low salt diet.
  Interventions: Other: Low Salt Diet; Other: Liberal salt diet
- Liberal salt/Low salt diet (Experimental): Cross-over trial of low salt and liberal salt diet
  Interventions: Other: Low Salt Diet; Other: Liberal salt diet

INTERVENTIONS:
Other: Low Salt Diet — On Day 0, patients will be randomized to one of the two crossover liberal/low or low/liberal salt diet groups. Each subject will complete two controlled dietary phases: 10-days of low salt diet, a washout period of 3-days, and 10-days of liberal salt diet.
Other: Liberal salt diet — On Day 0, patients will be randomized to one of the two crossover liberal/low or low/liberal salt diet groups. Each subject will complete two controlled dietary phases: 10-days of low salt diet, a washout period of 3-days, and 10-days of liberal salt diet.

SUMMARY:
The purpose of this study is to determine whether a salt restriction diet improves immune parameters in patients with autoimmune hepatitis.

DETAILED DESCRIPTION:
The etiology of autoimmune hepatitis (AIH) is unknown although both genetic and environmental factors are thought to be involved. A defect in immune regulation affecting regulatory T cells (Tregs) has been demonstrated in AIH. Tregs function in the maintenance of immune homeostasis by controlling autoreactive immune responses to self-antigens.

Rationale: the western diet has been postulated as a potential environmental risk factor for the increasing incidence of autoimmune diseases in developed countries. Data from the investigators' laboratory also suggests that increased dietary salt intake might represent an environmental risk factor for the development of autoimmune diseases through the induction of pathogenic Th17 cells. The dramatic in vitro effects of high salt on the induction of pathogenic Th17 cells from naïve human CD4 cells {Kleinewietfeld, Hafler. Nature. 2013 Apr 25;496(7446):518-22. doi: 10.1038/nature11868.}, and block of in vitro Treg suppression, in line with in vivo effects on worsening murine experimental autoimmune encephalomyelitis (EAE), have prompted the investigators to examine the effects of increased dietary sodium chloride in a human in vivo system.

The investigators hypothesize that excess dietary salt may function as an environmental trigger that favors induction and expansion of pathogenic Th17 cells and leads to functional impairment of Tregs, thereby favoring development of autoimmunity. The investigators aim to study their established in vitro model in humans by altering the salt intake in patients over a 20-day period.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-50 years of age
* Children 1-17 years of age
* ALT and/or ALP/GGT level > 2X upper limit of normal
* ANA or SMA >/= 1:40
* ANA or SMA >/= 1:80
* or LKM >/= 1:40
* or SLA positive
* IgG > upper limit of normal

Exclusion Criteria:

* Chronic hepatitis C
* Decompensated Liver Disease

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in production of pathogenic TH17 cells. | 26 days
  Measuring TH17 cells by flow cytometry and qRT-PCR. There are no known normal ranges. The investigator will calculate the change by observing the difference from baseline values.

SECONDARY OUTCOMES:
Change from baseline in regulatory T cell function. | 26 days
  Measuring T cell function by flow cytometry. There are no known normal ranges. The investigator will calculate the change by observing the difference from baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Udeme Ekong, MD, MPH, Principal Investigator — Yale University